CLINICAL TRIAL: NCT05370911
Title: Effects of Repeated Dosing of Psilocybin on Obsessive-Compulsive Disorder: A Randomized, Waitlist-Controlled Study
Brief Title: Effects of Repeated Psilocybin Dosing in OCD
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Steven & Alexandra Cohen Foundation (Other)
Responsible Party: Principal Investigator, Benjamin Kelmendi, MD, Assistant Professor of Psychiatry, Yale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2000032623
Record Dates: First submitted 2022-04-19; First posted 2022-05-12 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Psilocybin
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Psilocybin

STUDY DESIGN:
Intervention Model Description: In the study, participants will be randomized to receive either immediate treatment with two doses of oral psilocybin separated by one week (n = 15) or enter a waitlist control/delayed treatment group and receive the same treatment 7 weeks post-randomization (n = 15).
Who Masked: Outcomes Assessor
Masking Description: Only the independent rater for each participant will be blinded to their condition; blind will be broken at the end of week 7 (i.e., 4 weeks post-second dosing), after which participants in the waitlist/delayed treatment group will begin their treatment phase.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immediate Treatment (Experimental): Participants randomized to this condition will receive treatment immediately, facilitated by two study staff members, and which consists of two preparatory sessions, followed by the first dosing session and two integration sessions, then the second dosing session and two integration sessions. This is followed by follow-up and long-term follow-up visits up to 12 months post-second dose.
  Interventions: Drug: Psilocybin
- Waitlist Control/Delayed Treatment (No Intervention): Participants randomized to this condition will first enter a waitlist phase that lasts for 7 weeks, after which rater unblinding will occur, and participants will be rescreened. If participants remain eligible at this time, they will begin their treatment phase. During their treatment phase, participants in this condition will receive the same treatment as described for participants in the immediate treatment group. This is followed by follow-up and long-term follow-up visits up to 12 months post-second dose.

INTERVENTIONS:
Drug: Psilocybin — The first oral dose will be 25 mg, and the second dose will be either 25 mg or 30 mg, depending on response to first dose.
  Psilocybin is a naturally occurring hallucinogenic ingredient found in some varieties of mushrooms that can be produced synthetically. It is considered to be a serotonergic psychedelic. We will use synthetically produced oral psilocybin in this study.
  Other Names:
  "Magic Mushrooms"
  Arms: Immediate Treatment

SUMMARY:
This study aims to investigate the effects of repeated dosing of oral psilocybin on obsessive-compulsive disorder (OCD) symptomatology in a randomized, waitlist-controlled design with blinded independent ratings, and assess psychological mechanisms that may mediate psilocybin's therapeutic effects on OCD.

DETAILED DESCRIPTION:
Aim 1: To examine the effects of two doses of psilocybin on OCD symptoms among participants in the immediate treatment condition, compared to participants in the waitlist control/delayed treatment condition. The investigators hypothesize that participants in the immediate treatment group will report statistically significantly greater symptom improvement from baseline 4 days post-second dose, compared to participants in the waitlist control/delayed treatment group at the same interval during their waitlist phase.

Aim 2: To examine the effects of two doses of psilocybin on OCD symptoms, compared to one dose. The investigators hypothesize that two doses of oral psilocybin will reduce OCD symptoms to a statistically significantly greater extent than one dose.

This study aims to investigate the effects of repeated dosing of oral psilocybin on OCD symptomatology and assess psychological mechanisms that may mediate psilocybin's therapeutic effects on OCD. This study will employ a randomized, waitlist-controlled design with blinded independent ratings, with participants randomized to receive either immediate treatment (two doses oral psilocybin separated by one week) or delayed treatment (7 weeks post-randomization). An adaptive dose selection strategy will be implemented, with the first dose being standardized at 25 mg of psilocybin, and the second dose being either the same or a higher dosage (i.e., 30 mg) on the basis of a clinically significant response from baseline or not, respectively, 4 days post-first dose.

This study is conducted entirely on an outpatient basis with the possibility of remote/virtual follow-up visits after each dosing session. The dosing sessions last the entire day, and participants will be medically cleared prior to being permitted to return home with assistance (e.g., driven by a family member or friend, or ride share).

ELIGIBILITY:
Inclusion Criteria:

1. Primary DSM-5 diagnosis of OCD, with Y-BOCS-II score of 26 or greater at screening
2. Failed at least one medication and/or therapy trial of standard care treatment for OCD
3. English fluency
4. Agree to sign a medical release for investigators to communicate directly with participants' providers to confirm medication and psychotherapy histories or arrange contingencies in event of crises.
5. Agree to provide an adult contact (relative, spouse, close friend or other caregiver) who is willing and able to be reached by the PI and/or study personnel in the event of an emergency, and who can provide transportation for study visits and independently comment on any changes in the participant's mood or behavior after each administration of psilocybin.
6. Agree to commit to all study procedures.
7. Ability to orally ingest pills for psilocybin dosing visits.
8. Agree to adhere to lifestyle and medication modifications.
9. Must not be on psychotropic medications for OCD or comorbid psychiatric conditions for at least 8 weeks at the time of randomization, and agree to refrain from taking or starting any psychiatric medications until after 4 weeks post-second dose.
10. Must not be in current psychotherapy (CBT or ERP) and must not start new course of psychotherapy (CBT or ERP) for OCD or comorbid psychiatric conditions until after 4 weeks post-second dose.
11. If participant is of childbearing potential, must have a negative pregnancy test at study entry and prior to each dosing session.
12. If participant is of childbearing potential, agree to use adequate birth control and not attempt to become pregnant during study up to 4 weeks post-second dose.

Exclusion Criteria:

1. Personal or immediate (first-degree relative) family history of formally diagnosed schizophrenia or other psychotic disorders, or bipolar I/II disorder
2. Lack of knowledge about biological families' medical history, due to adoption or other circumstance
3. Active suicidal intent or suicidal or non-suicidal self-injurious behaviors
4. Unremitted Tourette syndrome
5. Lifetime diagnosis of autism spectrum disorder
6. Current substance use disorder (except for mild alcohol use disorder)
7. Any neurological condition, including history of seizure(s) or chronic/severe headaches
8. Any history of head injury with loss of consciousness for more than 30 min
9. Any use of classic psychedelic substances within the prior 12 months
10. Unwillingness to abstain from use of classic psychedelics outside of the study up to 4 weeks post-second dose.
11. Use of tobacco products or a THC-containing product more than 2 times per week on average over the past 30 days at screening.
12. Unwilingness or inability to abstain from use of tobacco or THC-containing products from 1 week prior to randomization up to 4 weeks post-second dose.
13. Positive urine drug test for any prohibited substance at screening or days of dosing, or positive breathalyzer test for alcohol on days of dosing
14. Unwillingness or inability to abstain from alcohol use at least 24 hours prior to the days of dosing, up to 24 hours after each dosing day (or corresponding intervals for waitlist group).
15. Any medical conditions that may render study procedures unsafe, including hypertension, history of cardiovascular disease, moderate-to-severe hepatic or renal impairment, diabetes, and hypo- or hyperthyroidism.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-07-20 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Change in Yale-Brown Obsessive-Compulsive Scale-Second Edition (Y-BOCS-II) Severity Scale total score from baseline at 4 days post-second dose | Baseline & 4 days post-second dose
  Clinician-administered assessment of severity of OCD symptoms over the past seven days. The most prominent obsessions and compulsions are rated on the Severity Scale from 0 to 4. Total Y-BOCS-II scores range from 0 to 40, with higher scores indicating greater severity of OCD symptoms.

SECONDARY OUTCOMES:
Change in Montgomery-Asberg Depression Scale (MADRS) total score from baseline at 4 days post-second dose | Baseline & 4 days post-second dose
  Clinician-administered assessment of severity of depressive symptoms over past month. Total scores range from 0 to 60, with higher scores indicating greater severity of depressive symptoms.
Change in Dimensional Obsessive-Compulsive Scale (DOCS) total score from baseline at 4 days post-second dose | Baseline & 4 days post-second dose
  Self-report measure of various OCD symptoms over the modified time frame of the past week. Total scores range from 0 to 140, with higher scores indicating greater severity of OCD symptoms.
Change in Obsessive Beliefs Questionnaire-44 (OBQ-44) total score from baseline at 4 days post-second dose | Baseline & 4 days post-second dose
  Self-report measure of various obsessive beliefs implicated in OCD in general. Total scores range from 44 to 308, with higher scores indicating greater severity of obsessive beliefs.
Change in Acceptance and Action Questionnaire for Obsessions and Compulsions (AAQ-OC) total score from baseline at 4 days post-second dose | Baseline & 4 days post-second dose
  Self-report measure of experiential avoidance and psychological flexibility in the context of OCD symptoms in general. Total scores range from 13 to 91, with higher scores indicating greater psychological inflexibility.
Change in Tolerance of Uncontrollability Questionnaire (TOUQ) total score from baseline at 4 days post-second dose | Baseline & 4 days post-second dose
  Self-report measure of ability to tolerate uncontrollability (or inversely need for control) in general. Total scores range from 19 to 133, with higher scores indicating greater tolerance of uncontrollability.
Change in White Bear Suppression Inventory (WBSI) total score from baseline at 4 days post-second dose | Baseline & 4 days post-second dose
  Self-report measure of thought suppression tendencies in general. Total scores range from 15 to 75, with higher scores indicating stronger thought suppression tendencies.
Change in Difficulties in Emotion Regulation Scale (DERS) total score from baseline at 4 days post-second dose | Baseline & 4 days post-second dose
  Self-report measure of emotion regulation difficulties in general. Total scores range from 36 to 180, with higher scores indicating greater difficulties with regulating emotions.
Change in Southampton Mindfulness Questionnaire (SMQ) total score from baseline at 4 days post-second dose | Baseline & 4 days post-second dose
  Self-report measure of trait mindfulness in regards to distressing thoughts and images. Total scores range from 0 to 96, with higher scores indicating greater trait mindfulness.
Toronto Mindfulness Scale (TMS) | Up to 3 weeks for immediate treatment condition, and up to 10 weeks for waitlist condition
  Self-report measure of state mindfulness during dosing session. Total scores range from 0 to 52, with higher scores indicating greater state mindfulness.
Set, Setting, and Intentions (SSI) Scale | Up to 3 weeks for immediate treatment condition, and up to 10 weeks for waitlist condition
  Self-report measure of set, setting, and clarity of intentions just prior to dosing session. Total mean scores range from 0 to 100 (after reverse-scoring two items), with higher scores indicating greater preparedness for the dosing session.
Mystical Experience Questionnaire (MEQ) | Up to 3 weeks for immediate treatment condition, and up to 10 weeks for waitlist condition
  Self-report measure of acute mystical experiences during dosing. Total mean scores range from 0 to 5, with higher scores indicating greater mystical experiences.
Psychological Insight Questionnaire (PIQ) | Up to 3 weeks for immediate treatment condition, and up to 10 weeks for waitlist condition
  Self-report measure of acute psychological insights during dosing. Total mean scores range from 0 to 5, with higher scores indicating greater insightful experiences.
Challenging Experience Questionnaire (CEQ) | Up to 3 weeks for immediate treatment condition, and up to 10 weeks for waitlist condition
  Self-report measure of acute challenging experiences during dosing. Total mean transformed scores range from 0 to 1, with higher scores indicating greater challenging experiences.
Ego Dissolution Inventory (EDI) | Up to 3 weeks for immediate treatment condition, and up to 10 weeks for waitlist condition
  Self-report measure of acute experiences of ego dissolution during dosing. Total mean scores range from 0 to 100, with higher scores indicating greater ego dissolution.
Emotional Breakthrough Inventory (EBI) | Up to 3 weeks for immediate treatment condition, and up to 10 weeks for waitlist condition
  Self-report measure of different experiences of emotional breakthroughs during dosing. Total mean scores range from 0 to 100, with higher scores indicating greater emotional breakthrough.
Change in Self-Compassion Scale (SCS) total mean score from baseline at 4 days post-second dose | Baseline & 4 days post-second dose
  Self-report measure of self-compassion in general. Total mean scores range from 1 to 5 (after reverse-scoring 13 items), with higher scores indicating greater self-compassion.
Change in Ten-Item Personality Inventory (TIPI) total score from baseline at 4 days post-second dose | Screening, 4 days and 12 months post-second dose
  Brief self-report measure of Big Five personality dimensions. Total scores range from 10 to 70 (after reverse-scoring 5 items), with higher scores indicating more positive personality traits.
Change in Persisting Effects Questionnaire (PEQ) subscale scores from 4 weeks post-second dose at 12 months post-second dose | 4 weeks post-second dose & 12 months post-second dose
  Self-report measure of persisting effects from dosing in general. Subscale scores range from a minimum of 0 to a maximum of 5 to 85, with higher scores indicating greater positive or negative persisting changes since dosing.
Change in Alcohol Use Disorders Identification Test (AUDIT) total score from baseline at 4 weeks post-second dose | Baseline & 4 weeks post-second dose
  Self-report measure of alcohol use severity. Total scores range from 0 to 40, with higher scores indicating greater alcohol use severity.
Change in Drug Use Disorders Identification Test (DUDIT) total score from baseline at 4 weeks post-second dose | Baseline & 4 weeks post-second dose
  Self-report measure of illicit substance use. Total scores range from 0 to 44, with higher scores indicating greater illicit substance use severity.
Change in Fagerstrom Test for Nicotine Dependence (FTND) total score from baseline at 4 weeks post-second dose | Baseline & 4 weeks post-second dose
  Self-report measure of nicotine use. Total scores range from 0 to 10, with higher scores indicating greater nicotine use severity.
Change in World Health Organization Disability Assessment Scale, v2.0 (WHODAS-2.0) 12-item, self-administered version total score from baseline at 4 days post-second dose | Baseline & 4 weeks post-second dose
  Self-report measure of symptom-related functional impairment in general. Total scores range from 12 to 60, with higher scores indicating greater functional impairment.
Change in Quality of Life Enjoyment & Satisfaction Questionnaire - Short Form (Q-LES-Q-SF) percentage maximum score from baseline at 4 days post-second dose | Baseline & 4 weeks post-second dose
  Self-report measure of life satisfaction over the past week. Percentage maximum scores range from 0% to 100%, with higher percentages indicating greater life satisfaction.
Writing task | Baseline & 4 days post-second dose
  Online writing task in which participants describe their perceptions of their OCD symptoms with a short written essay
Columbia Suicide Severity and Risk Scale (C-SSRS) Since Last Visit version | Every study visit through study completion, an average of 12 months and 3 weeks for immediate treatment condition, and an average of 12 months and 10 weeks for waitlist condition
  Clinician-administered assessment of suicidal ideation and behaviors since the last study visit
Theoretical Orientation Profile Scale-Revised (TOPS-R) | Baseline
  Clinician-reported measure of theoretical orientation over 11 subscales, each corresponding to a different theoretical orientation. Subscale scores range from 1 to 30, with higher scores indicating greater affiliation with a particular theoretical orientation.
Working Alliance Inventory-Short Revised (WAI-SR) | Up to 4 days post-second dose
  Self-report measure of perceived working alliance with study clinicians. Total scores range from 0 to 60, with higher scores indicating stronger perceived working alliance.
Change in Symptom Provocation Task (SPT) ratings from baseline at 4 days post-second dose | Baseline & 4 days post-second dose
  Behavioral measure of OCD symptoms when provoked with idiosyncratic questions. Scores for compulsive urges range from 0-10 in terms of VAS ratings, with higher VAS ratings indicating greater compulsive urges.
Stanford Expectations of Treatment Scale (SETS) | Baseline
  Self-report measure of treatment expectancy over 2 subscales, corresponding to positive and negative expectancy. Subscale scores range from 7 to 21, with higher scores indicating more positive or negative expectancy.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Kelmendi, MD, Principal Investigator — Yale University; Terence Ching, PhD, Principal Investigator — Yale University; Christopher Pittenger, MD, PhD, Study Director — Yale University
Locations (1):
- Yale OCD Research Clinic (40 Temple St, 4th Floor), New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moreno FA, Wiegand CB, Taitano EK, Delgado PL. Safety, tolerability, and efficacy of psilocybin in 9 patients with obsessive-compulsive disorder. J Clin Psychiatry. 2006 Nov;67(11):1735-40. doi: 10.4088/jcp.v67n1110. PMID 17196053
- [Background] Davis AK, Barrett FS, May DG, Cosimano MP, Sepeda ND, Johnson MW, Finan PH, Griffiths RR. Effects of Psilocybin-Assisted Therapy on Major Depressive Disorder: A Randomized Clinical Trial. JAMA Psychiatry. 2021 May 1;78(5):481-489. doi: 10.1001/jamapsychiatry.2020.3285. PMID 33146667
- [Background] Ross S, Bossis A, Guss J, Agin-Liebes G, Malone T, Cohen B, Mennenga SE, Belser A, Kalliontzi K, Babb J, Su Z, Corby P, Schmidt BL. Rapid and sustained symptom reduction following psilocybin treatment for anxiety and depression in patients with life-threatening cancer: a randomized controlled trial. J Psychopharmacol. 2016 Dec;30(12):1165-1180. doi: 10.1177/0269881116675512. PMID 27909164
- [Background] Griffiths RR, Johnson MW, Carducci MA, Umbricht A, Richards WA, Richards BD, Cosimano MP, Klinedinst MA. Psilocybin produces substantial and sustained decreases in depression and anxiety in patients with life-threatening cancer: A randomized double-blind trial. J Psychopharmacol. 2016 Dec;30(12):1181-1197. doi: 10.1177/0269881116675513. PMID 27909165
- [Derived] Ching THW, Amoroso L, Bohner C, D'Amico E, Eilbott J, Entezar T, Fitzpatrick M, Fram G, Grazioplene R, Hokanson J, Kichuk SA, Martins B, Patel P, Schaer H, Shnayder S, Witherow C, Pittenger C, Kelmendi B. Safety, feasibility, tolerability, and clinical effects of repeated psilocybin dosing combined with non-directive support in the treatment of obsessive-compulsive disorder: protocol for a randomized, waitlist-controlled trial with blinded ratings. Front Psychiatry. 2024 Jan 9;14:1278823. doi: 10.3389/fpsyt.2023.1278823. eCollection 2023. PMID 38264632